CLINICAL TRIAL: NCT03140605
Title: Hellenic Registry for Familial Hypercholesterolemia
Brief Title: Greek Registry - Familial Hypercholesterolaemia
Acronym: GRegistry-FH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hellenic College of Treatment of Atherosclerosis (Other)
Responsible Party: Principal Investigator, Genovefa Kolovou, M.D., Ph.D., F.E.S.C., S.F.S.A, Cardiologist, Head of Hellenic College of Treatment of Atherosclerosis, Hellenic College of Treatment of Atherosclerosis
Other Study IDs: 2017-HPLS-IIS
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Familial hypercholesterolemia (FH) [heterozygous (heFH) or homozygous FH (hoFH)] is a common genetic disorder, characterized by elevated plasma low density lipoprotein (LDL) cholesterol concentration leading (if untreated) to cholesterol deposits in the corneas, eyelids and extensor tendons, rapidly progressing vascular disease, and aortic valve disease.

DETAILED DESCRIPTION:
In contrast, timely recognition and effective treatment of FH can result in a significant improvement in clinical outcomes. The problem is that that majority of individuals with FH are unaware of their disease, particularly that the disease remains silent for many years. In most countries around the world <5% of individuals with FH are identified .

Until lately the prevalence of heFH was traditionally considered to be ~ 1:500 individuals , although clinical and genetic studies suggest that heFH affects ~ 1:200-250 individuals . Thus, the aim of the Hellenic College of Treatment of Atherosclerosis (HCAT) is to 1). Evaluate the prevalence of FH in Greece (FHG-Registry) and 2). To inform population of FH disease.

ELIGIBILITY:
Inclusion Criteria:

* both genders
* >18 years, <80 years
* door to door enrolment
* eligible to sign informed consent

Exclusion Criteria:

* <18 years, >80 years
* deny to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample of citizents on Panhellenic basis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2020-12-10 (Estimated); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
the prevalence of Familiar Hypercholesterolaemia in Greece | 1 month
  patients with FH will be screened and include in Registry

CONTACTS AND LOCATIONS:
Locations (1):
- Onassis Cardiology Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kolovou GD, Damaskos DS, Anagnostopoulou KK, Salpea KD, Dritsas A, Giannakopoulou V, Vasiliadis IK, Cokkinos DV. Stress testing response in women heterozygous for familial hypercholesterolemia. Int J Cardiol. 2007 Oct 31;122(1):96-7. doi: 10.1016/j.ijcard.2006.11.046. Epub 2007 Jan 18. PMID 17239976
- [Background] Kolovou GD, Dedoussis GV, Anagnostopoulou KK, Hatzigeorgiou GCh, Salpea KD, Choumerianou DM, Rammos S, Mikhailidis DP, Cokkinos DV. Management of a patient with a null low-density lipoprotein receptor mutation: a case report. Angiology. 2006 Dec-2007 Jan;57(6):729-32. doi: 10.1177/0003319706294421. PMID 17235114
- [Background] Kolovou GD, Kostakou PM, Anagnostopoulou KK. Familial hypercholesterolemia and triglyceride metabolism. Int J Cardiol. 2011 Mar 17;147(3):349-58. doi: 10.1016/j.ijcard.2010.08.009. Epub 2010 Sep 9. PMID 20826022
- [Background] Markousis-Mavrogenis G, Mavrogeni S, Kolovou G. Early coronary artery disease--Usual and unusual suspects. Int J Cardiol. 2016 Jan 1;202:511. doi: 10.1016/j.ijcard.2015.09.050. Epub 2015 Sep 25. No abstract available. PMID 26447655
- [Background] Beliard S, Millier A, Carreau V, Carrie A, Moulin P, Fredenrich A, Farnier M, Luc G, Rosenbaum D, Toumi M, Bruckert E; French FH Registry group. The very high cardiovascular risk in heterozygous familial hypercholesterolemia: Analysis of 734 French patients. J Clin Lipidol. 2016 Sep-Oct;10(5):1129-1136.e3. doi: 10.1016/j.jacl.2016.06.007. Epub 2016 Jun 27. PMID 27678429
- [Background] Mundal L, Igland J, Ose L, Holven KB, Veierod MB, Leren TP, Retterstol K. Cardiovascular disease mortality in patients with genetically verified familial hypercholesterolemia in Norway during 1992-2013. Eur J Prev Cardiol. 2017 Jan;24(2):137-144. doi: 10.1177/2047487316676135. Epub 2016 Oct 28. PMID 27794106
- [Background] EAS Familial Hypercholesterolaemia Studies Collaboration; Vallejo-Vaz AJ, Akram A, Kondapally Seshasai SR, Cole D, Watts GF, Hovingh GK, Kastelein JJ, Mata P, Raal FJ, Santos RD, Soran H, Freiberger T, Abifadel M, Aguilar-Salinas CA, Alnouri F, Alonso R, Al-Rasadi K, Banach M, Bogsrud MP, Bourbon M, Bruckert E, Car J, Ceska R, Corral P, Descamps O, Dieplinger H, Do CT, Durst R, Ezhov MV, Fras Z, Gaita D, Gaspar IM, Genest J, Harada-Shiba M, Jiang L, Kayikcioglu M, Lam CS, Latkovskis G, Laufs U, Liberopoulos E, Lin J, Lin N, Maher V, Majano N, Marais AD, Marz W, Mirrakhimov E, Miserez AR, Mitchenko O, Nawawi H, Nilsson L, Nordestgaard BG, Paragh G, Petrulioniene Z, Pojskic B, Reiner Z, Sahebkar A, Santos LE, Schunkert H, Shehab A, Slimane MN, Stoll M, Su TC, Susekov A, Tilney M, Tomlinson B, Tselepis AD, Vohnout B, Widen E, Yamashita S, Catapano AL, Ray KK. Pooling and expanding registries of familial hypercholesterolaemia to assess gaps in care and improve disease management and outcomes: Rationale and design of the global EAS Familial Hypercholesterolaemia Studies Collaboration. Atheroscler Suppl. 2016 Dec;22:1-32. doi: 10.1016/j.atherosclerosissup.2016.10.001. Epub 2016 Dec 7. PMID 27939304
- [Derived] Kolovou G, Makrygiannis S, Marvaki C, Pavlatou N, Anagnostopoulou K, Giannakopoulou V, Goumas G, Kalogeropoulos P, Kolovou V, Limberi S, Perrea D, Tzenalis A, Emre Z, Jahaj E, Kasiara Z, Giannakoulis I, Tsolakoglou I, Kadda O, Tsaloukidis N, Koulaxidou R, Marvaki A, Foussas S, Melidonis A, Hoursalas G, Vlachopoulos C, Katsiki N, Milionis H, Liberopoulos E, Bilianou H. Prevalence and Risk Factors for Atherosclerotic Cardiovascular Disease in 7704 Individuals: An Analysis from the Greek Registry for the Prevalence of Familial Hypercholesterolemia (GRegistry-FH). J Cardiovasc Dev Dis. 2024 Dec 23;11(12):411. doi: 10.3390/jcdd11120411. PMID 39728301